CLINICAL TRIAL: NCT03945916
Title: The Effect of Dark Chocolate on Metabolism and Performance in Trained Cyclists at Simulated Altitude
Brief Title: Dark Chocolate and Exercise Performance in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 189
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Crossover - dark chocolate vs. placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dark chocolate (Experimental): 180g/d dark chocolate
  Interventions: Dietary Supplement: Dark chocolate
- Placebo (Placebo Comparator): 180g/d of artificial dark chocolate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dark chocolate — 180 g/d dark chocolate for 15 days followed by exercise testing
  Arms: Dark chocolate
Dietary Supplement: Placebo — Placebo: 180 g/d imitation dark chocolate for 15 days followed by exercise testing
  Arms: Placebo

SUMMARY:
Nitrate supplements (beetroot juice, pure sodium nitrate) have become common among endurance athletes because the ingestion of exogenous nitrate leads to increased levels of nitric oxide (NO) in the body. Increased NO has been shown to have various performance enhancing effects such as increased muscle contractility, increased blood flow through vasodilation, mitochondrial biogenesis, and improved glucose uptake. Supplementation with exogenous forms of nitrate has also been shown to improve cycling performance in the oxygen deprived environment of simulated altitude through increased muscular oxygenation. Further research is emerging that suggests that dark chocolate (DC) may have similar effects through flavonoids, a bioactive micronutrient that increases the synthesis of NO and reduces the rate at which NO is removed from the blood. In addition to performance enhancement, the flavonoids in DC also have anti-inflammatory and antioxidant effects, which could reduce muscle damage after a bout of exercise and increase the rate at which the muscle recovers. The purpose of this research is to investigate the effects of DC on cycling performance and recovery in cyclists at altitude. it is hypothesised that the DC condition will result in superior metabolism during exercise and increase muscular oxygenation, leading to improved performance while enhancing recovery from exercise.

Methods: 12 trained cyclists will be randomized to supplement with 160g of DC or an isocaloric placebo per day for 2 weeks in a cross-over study. After the 2-weeks of supplementation participants will attend a lab session in which they will cycle 90 minutes at 60% VO2max followed immediately by a 10km time trial (TT) at a simulated altitude of 1500m (15% O2). Plasma levels of blood glucose and lactate will be measured before, throughout, and after exercise while muscular and cerebral oxygenation will be measured continuously throughout exercise. Recovery of the knee extensors will be assessed before and immediately after exercise as well as 24 and 48 hours later by determining knee extensor strength and muscle pain.

DETAILED DESCRIPTION:
Dark chocolate is rich in flavonoids, bioactive micronutrients that increase the bioavailability of nitric oxide as well as decrease the rate in which nitric oxide is removed from the body. Through increasing the bioavailability of nitric oxide (NO) to bodily tissues, the tissues are better able to utilize oxygen, synthesize energy, and utilize glucose from the blood. In addition to increasing the bioavailability of nitric oxide, the flavonoids in dark chocolate also have antioxidant properties, which reduce oxidative stress and inflammation in the muscle. These anti-inflammatory and antioxidant properties have been show to alleviate muscle damage after intense exercise and improve recovery. These factors are of benefit for endurance athletes through improving performance and enhancing recovery from exercise.

Studies investigating the effects of dark chocolate on exercise performance are few, and thus more research is needed to strengthen evidence for or against dark chocolate for endurance exercise performance. Dark chocolate has been shown to improve time trial performance in some studies due to the increased bioavailability of NO while showing no effect on performance in others, displaying an inconsistency in the literature. Although oxidative stress has been studied, no studies to date have investigated the effects of dark chocolate on the product of this stress, muscle damage. To measure muscular damage, we will be assessing muscular pain and force recovery.

Dark chocolate also contains caffeine and theobromine (73mg and 883mg per 100g serving, respectively) Caffeine and theobromine have been shown to have beneficial effects on exercise performance through increasing fatty acid mobilization and slowing the onset of fatigue.

Finally, carbohydrates with a low glycemic index are better than those with a high glycemic index for stimulating fat usage at the muscle and therefore have potential to improve endurance exercise performance because endurance performance is limited by carbohydrate availability in the muscle. Dark chocolate has a glycemic index of 23, meaning it has very little effect on blood sugar, and thus results in lower insulin release than other carbohydrates (insulin inhibits fat usage at the muscle). Thus, dark chocolate may have performance enhancing effects through the mechanisms of nitric oxide, caffeine, and theobromine while providing carbohydrates that cause a reduced spike in blood sugar compared to other carbohydrate sources often used by athletes such as energy bars and gels.

In the current study the investigators are testing the effects of dark chocolate on cycling at altitude because some of the most important cycling races (e.g. Tour de France) involve cycling through mountain stages. Altitude places an extra challenge on cyclist because of the lower partial pressure of oxygen in the atmosphere. A food such as chocolate, which is proposed to enhance oxygen deliver to muscle may be ideal for exercise at altitude.

The research design is a double-blind cross-over study comparing two substances - dark chocolate and placebo (an artificial dark chocolate lacking cocoa-liquor). Participants will be randomized to one condition and then cross-over to the other condition after a one-month washout.

12 participants with consistent cycling experience will be recruited for this study. There will be 9 study visits.

Visit #1 will consist of testing maximal oxygen uptake (i.e. aerobic capacity) via a progressive cycling exercise test at normoxia (i.e. 20.93% O2) to determine eligibility for the study (the study includes only trained cyclists). The aerobic capacity test involves pedalling on a stationary bike with resistance increasing every minute until volitional fatigue. The test takes about 10-15 minutes (longer if the individual is of higher fitness). During the test, oxygen consumption is measured through a mouthpiece and the level of oxygen consumption is used as a measure of aerobic fitness. Participants will be deemed eligible if their maximal oxygen consumption is >50 ml/kg/min for males and >45 ml/kg/min for females.

Visit #2 will occur at least 3 days later and will consist of testing for ratings of muscle soreness (done at rest and by applying pressure to the quadriceps muscle using an algometer; i.e. a pressure gauge), maximal voluntary isometric contraction of the knee extensor muscle group, and aerobic capacity on a cycle ergometer at a simulated altitude of 2500m (15% O2) to determine workload to be used for subsequent testing. Visit #2 will also include a practice of a 10 km time trial on a cycle ergometer, which will be the performance indicator in the dark chocolate testing. During the 10 km time trial, the cyclist attempts to complete 10 km as fast as possible on a stationary bike.

Visit #3 will consist of a familiarisation trial using the actual cycling protocol used in the study (i.e. 90 minutes of cycling at an intensity corresponding to 60% maximal oxygen uptake reached during the aerobic capacity test in visit #2 plus a 10 km time trial, all at simulated altitude). The familiarisation trial is necessary to reduce the amount of variability across subsequent testing sessions (i.e. the subsequent testing sessions which compare dark chocolate to a control chocolate).

After visit #3, participants will be randomised to receive dark chocolate or a dark chocolate placebo. This will be consumed twice a day (160 g/d) for 14 days to deliver an appropriate dose of flavonoids in the dark chocolate condition to reduce inflammation and oxidation and have the desired effect on the endothelium of the blood vessels for release of nitric oxide. The amount of calories/carbohydrate to be consumed in the dark chocolate condition will be matched to the placebo control chocolate. Two days before visit #4 (i.e. on the 13th and 14th day of chocolate supplementation) participants will be instructed to try to minimise the amount of polyphenols they consume in their diet by minimising intake of fruits, vegetables, tea, coffee, alcohol, chocolate, cereals, wholemeal bread, and grains. Participants will keep food diaries by recording all foods and drinks they consume for these two days. These diaries will be photocopied and given back for the testing of the opposite chocolate condition in the next phase.

Visit #4 will occur on the 15th day of chocolate supplementation. Participants will come into the lab after an overnight fast (at least 10 hours). Reactivity of the blood vessels will be assessed using flow mediated dilation, a method in which the brachial artery in the arm is occluded for 5 minutes using a blood pressure cuff and the diameter of the artery is measured during occlusion as well as upon release of the cuff via ultrasound to assess how the blood vessel responds. They will then be tested again for muscle soreness, and maximal isometric voluntary contraction. They will be given 80 g dark chocolate or placebo and will sit quietly for 60 minutes prior to exercise testing. The timing and dose of the chocolate are to optimise carbohydrate availability prior to exercise and because the bio-availability of epicatechin (the main flavonoid in dark chocolate) peaks between 90-150 minutes post-ingestion, a time that would coincide with the exercise testing. The exercise testing will involve 90 minutes of cycling at a simulated altitude of 2500 m (15% O2) at 60% the aerobic capacity reached on the aerobic capacity test at simulated altitude (visit #2), followed by a 10 km time trial, also at altitude, where participants will cover 10 km as fast as they can. The total amount of time for this test (i.e. approximately 105 minutes) was chosen because recovery from cycling tests of this duration benefit from other forms of antioxidant rich substances such as cherry juice. After the time trial, muscle soreness, maximal voluntary contraction will be determined.

Visit #5 to the lab will occur the next morning, again in a fasted state, to test recovery of muscle damage. Thirty minutes after consumption of a 80 g dose of the dark chocolate or calorie/carbohydrate-matched dark chocolate placebo, muscle soreness, and maximal voluntary contraction will be determined. Participants will consume 80 g of the dark chocolate or dark chocolate flavoured placebo before bedtime. Visit #6 will occur the next morning and involve the same procedures as visit #5 (again to test recovery of muscle damage).

Visits 7, 8, and 9 will occur a month later after 14 days dark chocolate or dark chocolate flavoured placebo control supplementation (i.e. the opposite condition to what the participant received prior to visit #4). All testing will be identical to tests in visits #4, 5, and 6. A month between conditions was chosen to allow more than adequate wash- out of flavonoids from the dark chocolate and to ensure that any females who participate in the study are doing the exercise testing at approximately the same phase of their menstrual cycle because hormone fluctuations during the menstrual cycle can have a small impact on exercise performance.

The 10 km time trial performance will be assessed with a one-factor repeated measures ANOVA to compare dark chocolate vs. dark chocolate flavoured placebo. The recovery of strength (muscle damage) will be assessed with a 2-factor repeated measures ANOVA with factors of condition (dark vs. dark chocolate flavoured palcebo) and time (before, after, 1 day after, and 2 days after exercise).

Secondary endpoints include fat and carbohydrate oxidation during the exercise test, rating of perceived exertion, blood glucose and lactate, l and flow mediated dilation. All will be assessed with a chocolate x time repeated measures ANOVA

ELIGIBILITY:
Inclusion Criteria:

* Endurance-trained cyclists

Exclusion Criteria:

* Regular consumption of dark chocolate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
10 km time trial performance | Measured on day 15 of dark chocolate/placebo consumption
  cycling exercise performance

SECONDARY OUTCOMES:
Glucose | Change from baseline to 90 minutes of exercise
  Glucose during exercise
Lactate | Change from baseline to 90 minutes of exercise
  lactate during exercise
Muscle oxygenation | Change from baseline to 90 minutes of exercise
  Muscle oxygenation during exercise
Carbohydrate oxidation | Change from baseline to 90 minutes of exercise
  carbohydrate oxidation during exercise
Fat oxidation | Change from baseline to 90 minutes of exercise
  fat oxidation during exercise
Muscle soreness | Change from baseline to immediately after and 24 and 48 hours after exercise
  Assessment of post-exercise muscle soreness. This is done by applying 20 kg pressure with an algometer to the thigh and asking the participant to rate their soreness on a scale of 0 (no soreness) to 100 (worst soreness)
Muscular strength | Change from baseline to immediately after and 24 and 48 hours after exercise
  Maximal voluntary contraction

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - University of Regain, Faculty if Kinesiology and Health Sciences, Regina, Saskatchewan
  - College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan